CLINICAL TRIAL: NCT01499264
Title: Efficacy of MySkin Patch for the Healing of Burn Wounds: a Randomised Controlled Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associazione Infermieristica per lo studio delle Lesioni Cutanee (Other)
Collaborators: Artsana S.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AISLeC-002
Record Dates: First submitted 2011-12-20; First posted 2011-12-26 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Burns; Burn Injury; Hydrogel Bandage; Occlusive Dressings
Keywords: MySkin patch
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MySkin patch (Experimental): Hydrogel e polyurethane film
  Interventions: Device: MySkin patch
- Traditional Dressing (Active Comparator)
  Interventions: Device: Traditional Dressing

INTERVENTIONS:
Device: MySkin patch — Hydrogel and polyurethane film
  Arms: MySkin patch
Device: Traditional Dressing — Gauze and Patch
  Arms: Traditional Dressing

SUMMARY:
Evaluation of clinical efficacy of my skin (hydrogel and polyurethane film) plus best practice clinical care in subjects with burn injuries with particular regard to: 1) Wound healing (complete reepithelialization), 2) the patient's pain. In the context of the study will be collected secondary outcomes related to type of lesion and its clinical evolution through the analysis of the items in the scale of the PSST.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one injury burn covered by a dressing of 10x8 cm (80 cm2)
* Injury treated with medication in use at the center
* Patients assisted at the emergency care, or at the outpatient
* Extension of the lesion less than 80 cm2 (including dressings in cm10x8cm)
* Patient age greater than or equal to 18 years
* Patients who have given consent to enrollment in the trial and the processing of personal data
* Patient / lesion that has already been recruited in the study or who have previously passed a period of 10 days (washout) of "no treatment" according to the research protocol

Exclusion Criteria:

* A end-stage of disease
* Suspected or known allergic diathesis to the product of medication
* Subjects that do not give consent to data processing
* Dry lesion with necrosis or eschar
* Presence of both local and systemic infection or inflammation
* Injuries that to the decision of the provider of care, needs a targeted local treatment other than as provided for in the Protocol
* Patient / lesion that has already been previously recruited into the study, before a period of 10 days (washout) of suspension from the same research protocol
* Patients who use alternative medicine treatments such as aloe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Wound healing and Significant reduction in pain | 1 month

SECONDARY OUTCOMES:
Clinical evaluation of the lesion scores for each visit, the presence / absence of infection for each visit | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia Tomasin, Study Director — Associazione Infermieristica per lo studio delle Lesioni Cutanee
Locations (2):
- Italy (2):
  - Istituto Clinico Humanitas - IRCCS, Rozzano, Milano
  - Ospedale di Circolo di Busto Arsizio, Busto Arsizio, Varese